CLINICAL TRIAL: NCT00459407
Title: Phase Ib Study of Polyphenon E in a Pre-prostatectomy Prostate Cancer Cohort
Brief Title: Defined Green Tea Catechins in Treating Patients With Prostate Cancer Undergoing Surgery to Remove the Prostate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2009-00894; HSC # 06-0695-04; N01CN35158 (NIH); CDR0000538554 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2013-02

CONDITIONS: Adenocarcinoma of the Prostate; Stage I Prostate Cancer; Stage II Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — polyphenon E; Immunohistochemistry; Immunoenzyme Techniques; Biopsy; Mass Spectrometry; Chromatography, High Pressure Liquid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (green tea catechin extract) (Experimental): Patients receive oral defined green tea catechin extract daily for 4-7 weeks.
  All patients undergo surgery one day after the last dose of study agent.
  Interventions: Dietary Supplement: defined green tea catechin extract; Other: immunohistochemistry staining method; Other: immunoenzyme technique; Other: laboratory biomarker analysis; Procedure: biopsy; Other: mass spectrometry; Other: high performance liquid chromatography
- Arm II (placebo) (Placebo Comparator): Patients receive oral placebo daily for 4-7 weeks.
  All patients undergo surgery one day after the last dose of study agent.
  Interventions: Drug: placebo; Other: immunohistochemistry staining method; Other: immunoenzyme technique; Other: laboratory biomarker analysis; Procedure: biopsy; Other: mass spectrometry; Other: high performance liquid chromatography

INTERVENTIONS:
Dietary Supplement: defined green tea catechin extract — Given orally
  Other Names: Polyphenon E
  Arms: Arm I (green tea catechin extract)
Drug: placebo — Given orally
  Other Names: PLCB
  Arms: Arm II (placebo)
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Other: immunoenzyme technique — Correlative studies
  Other Names: immunoenzyme techniques
Other: laboratory biomarker analysis — Correlative studies
Procedure: biopsy — Undergo biopsy
  Other Names: biopsies
Other: mass spectrometry — Correlative studies
Other: high performance liquid chromatography — Correlative studies
  Other Names: HPLC

SUMMARY:
Green tea extract contains ingredients that may prevent or slow the growth of prostate cancer. This phase I trial is studying how well green tea extract works in treating patients with prostate cancer undergoing surgery to remove the prostate

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the bioavailability of defined green tea catechin extract in prostate tissue after treatment with defined green tea extract in patients with prostate cancer.

SECONDARY OBJECTIVES:

I. Determine the effect of this treatment on changes in clusterin levels and matrix metalloproteinase (MMP)-2 and MMP-9 in prostate tissue from these patients.

II. Determine the effect of this treatment on changes in serum insulin-like growth factor (IGF)-1 and IGF binding protein-3 in these patients.

III. Determine the effect of this treatment on changes in oxidative DNA damage in peripheral blood leukocytes in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive oral defined green tea catechin extract daily for 4-7 weeks.

Arm II: Patients receive oral placebo daily for 4-7 weeks.

All patients undergo surgery one day after the last dose of study agent.

Biopsies are taken at the time of surgery. Plasma and tissue catechin levels are measured with high performance liquid chromatography (HPLC). 8OHdG levels in peripheral blood are measured with HPLC and mass spectometry. Immunohistochemistry is used to measure matrix metalloproteinase (MMP)-2, MMP-9, and clusterin. Insulin-like growth factor (IGF)-1 and IGF binding protein-3 are measured with immunoenzyme techniques.

ELIGIBILITY:
Criteria:

* Biopsy-proven adenocarcinoma of the prostate meeting the following criteria: organ-confined disease; treatable by prostatectomy
* PSA < 50 ng/mL
* ECOG performance status (PS) 0-1 or Karnofsky PS 70-100%
* Bilirubin normal
* AST and ALT normal
* Creatinine normal
* Fertile patients must use effective contraception
* No uncontrolled intercurrent illness including, but not limited to, any of the following: ongoing or active infection; symptomatic congestive heart failure; unstable angina pectoris; cardiac arrhythmia; psychiatric illness or social situations that would limit study compliance
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to green tea extract
* No prior therapy for prostate cancer (i.e., hormone therapy, radiation therapy, or surgery)
* No systemic treatment (chemotherapy) and/or radiation therapy for any malignancy within the past 5 years (excluding nonmelanoma skin cancer or cancer confined to organs with surgical removal as the only treatment)
* No regular tea consumption (> 6 servings of hot tea or 12 servings of iced tea or equivalent combination per week) within the past month
* No other concurrent investigational agents
* No other concurrent consumption of tea or tea-derived products from green, black, or oolong tea

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Post-treatment green tea catechin concentration levels in prostate tissue | Up to 6 weeks
  Descriptive statistics will be performed on prostate tissue EGCG within each intervention group. The difference in concentration levels between the two intervention groups will be tested using a two-group t-test at a one-sided 0.05 level of significance. If the distributions are not symmetrical, a non-parametric Wilcoxon test will be considered. The percentage of patients positive for EGCG in prostate tissue will be compared between the intervention groups using a Fisher's exact test of proportions at a one-sided 0.05 level of significance.

SECONDARY OUTCOMES:
Changes in clusterin, matrix metalloproteinase (MMP)-2, and MMP-9 levels | Baseline to post-treatment
  Will be compared between intervention groups using a two-group t-test with a 0.05 two-sided significance level; with a sample size of 23 patients per group, there will be over 90% power to detect a difference equal to an effect size of 1.0. If the distributions are not symmetrical, a non-parametric Wilcoxon test will be considered. Correlations among the various biomarkers, as well as between post-intervention EGCG concentrations and changes in biomarker levels, will be explored (using Pearson or Spearman Rank correlation coefficients as appropriate).
Changes in Serum levels of insulin-like growth factor (IGF)-1 and IGF binding protein-3 | Baseline to post-treatment
  Will be compared between intervention groups using a two-group t-test with a 0.05 two-sided significance level; with a sample size of 23 patients per group, there will be over 90% power to detect a difference equal to an effect size of 1.0. If the distributions are not symmetrical, a non-parametric Wilcoxon test will be considered. Correlations among the various biomarkers, as well as between post-intervention EGCG concentrations and changes in biomarker levels, will be explored (using Pearson or Spearman Rank correlation coefficients as appropriate).
Change in ratio of 8OHdG:dG | Baseline to post-treatment
  Statistical analysis will focus on the change scores (defined as changes from baseline to post-intervention). Changes in the Polyphenon E group will be compared with those in the placebo group, using a two-sided t-test.
Change in plasma levels of EGCG | Baseline to post-treatment
  Will be compared between groups, and the correlation of plasma and prostate tissue levels will be examined; however, plasma levels are expected to be low because of the washout during pre-operative fasting. Additional exploratory analyses will investigate the correlation of EGCG tissue levels with adherence during the intervention period (assessed primarily by capsule counts).

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Ahmann, Principal Investigator — Arizona Cancer Center - Tucson
Locations (1):
- Arizona Cancer Center - Tucson, Tucson, Arizona, United States

REFERENCES:
- [Derived] Nguyen MM, Ahmann FR, Nagle RB, Hsu CH, Tangrea JA, Parnes HL, Sokoloff MH, Gretzer MB, Chow HH. Randomized, double-blind, placebo-controlled trial of polyphenon E in prostate cancer patients before prostatectomy: evaluation of potential chemopreventive activities. Cancer Prev Res (Phila). 2012 Feb;5(2):290-8. doi: 10.1158/1940-6207.CAPR-11-0306. Epub 2011 Nov 1. PMID 22044694